CLINICAL TRIAL: NCT04880187
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study to Evaluate the Safety, Tolerability, and Efficacy of AXA1125 in Subjects With Non Cirrhotic, Non Alcoholic Steatohepatitis and Fibrosis (EMMPACT)
Brief Title: Safety, Tolerability, and Efficacy of AXA1125 in NASH With Fibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXA1125-101
Record Dates: First submitted 2021-05-03; First posted 2021-05-10 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-05

CONDITIONS: Non Alcoholic Steatohepatitis (NASH)
Keywords: Steatosis; Lobular inflammation; Ballooning; Liver biopsy; Liver fat; Liver stiffness; NASH; Aminio Acids; Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Fibrosis | interventions — leucine, isoleucine, valine, arginine, glutamine, and N-acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AXA1125 22.6g (Experimental): 22.6 g AXA1125 administered orally BID with or without food
  Interventions: Drug: AXA1125
- AXA1125 33.9g (Experimental): 33.9 g AXA1125 administered orally BID with or without food
  Interventions: Drug: AXA1125
- Placebo (Placebo Comparator): Matching Placebo administered orally BID with or without food
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXA1125 — AXA1125 administered BID with or without food
  Arms: AXA1125 22.6g; AXA1125 33.9g
Drug: Placebo — Matching Placebo administered BID with or without food
  Arms: Placebo

SUMMARY:
This study will compare the effects of AXA1125, an orally active mixture of amino acids, compared to placebo, on improving fat and inflammation (steatohepatitis) as well as fibrosis in subjects with non alcoholic steatohepatitis (NASH). as well as the safety and tolerability of AXA1125. Subjects will take one of two different doses of AXA1125 or a placebo twice daily, and a liver biopsy will be done at the beginning and end of the 48-week study.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and provide written informed consent.
* Male and female adults aged > 18 years.
* Must have NASH and fibrosis on a liver biopsy sample
* If a historical liver biopsy is used for Screening, obtained within 6 months prior to Screening;
* Subjects may have a diagnosis of T2DM

Exclusion Criteria:

* History or presence of liver disease (other than NAFLD or NASH)
* History or presence of cirrhosis and/or history or presence of hepatic decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in steatohepatitis | Baseline to Week 48
  2-point improvement from baseline to Week 48 in the non-alcoholic fatty liver disease (NAFLD) Activity Score (NAS) based on a scale from 0-8 with 0 being no NASH and 8 being the highest score

SECONDARY OUTCOMES:
Resolution of NASH without worsening of fibrosis | Baseline to week 48
  The proportion of subjects with resolution of NASH with no worsening of fibrosis defined as a post-treatment ballooning score of 0 and an inflammation score of 0 or 1 on liver biopsy.
Improvement of fibrosis by one stage without worsening of NASH | Baseline to week 48
  The proportion of subjects who have at least a 1-stage improvement in fibrosis and no worsening of NASH based on liver biopsy 0 being no fibrosis and 4 being the worse.
Incidence of study drug emergent adverse events (AEs) and serious adverse events (SAEs) | Baseline to week 48
Change from baseline in liver stiffness as measured by vibration controlled transient elastography (Fibroscan™) | Baseline to week 48
Change from baseline in hepatic fat as measured by MRI | Baseline to week 48
Change from baseline in measures of glucose control as determined by glycated hemoglobin (HbA1c) | Baseline to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Principal Investigator — Pinnacle Clinical Research
Locations (75):
- United States (57):
  - Cullman Clinical Trials, Cullman, Alabama
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - San Fernando Valley Health Institute, Canoga Park, California
  - National Research Institute, Gardena, California
  - National Research Institute, Huntington Park, California
  - OM Research LLC, Lancaster, California
  - National Research Institute, Los Angeles, California
  - Inland Empire Liver Foundation, Rialto, California
  - Precision Research Institute, LLC, San Diego, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Synergy Healthcare, Bradenton, Florida
  - Tampa Bay Medical Research , Inc., Clearwater, Florida
  - Evolution Clinical Trials, Inc., Hialeah Gardens, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - ENCORE Borland Groover Clinical Research, Jacksonville, Florida
  - ClinCloud LLC, Maitland, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - La Salud Research, Miami, Florida
  - Genoma Research Group, Inc, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Theia Clinical Research, LLC, Pinellas Park, Florida
  - Progressive Medical Research, Port Orange, Florida
  - ClinCloud, LLC, Viera, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - ASHA Clinical Research, Hammond, Indiana
  - Indiana University (IU) School of Medicine, Indianapolis, Indiana
  - Delta Research Partners, Bastrop, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Tandem Clinical Research GI, Metairie, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - The National Diabetes & Obesity Research Institute, Biloxi, Mississippi
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Sierra Clinical Research, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Tandem Clinical Research GI, New York, New York
  - Lucas Research - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Rapid City Medical Center, Rapid City, South Dakota
  - ClinSearch LLC, Chattanooga, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - American Research Corporation, Austin, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - R & H Clinical Research, Katy, Texas
  - EPIC Medical Research, Red Oak, Texas
  - American Research Corporation, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - R & H Clinical Research, Stafford, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Impact Clinical Research, Waco, Texas
  - Velocity - Advanced Clinical Research - Salt Lake City of Gastroenterolog, Riverton, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - Virginia Commonwealth University Medical College of Virginia, Richmond, Virginia
- Australia (5):
  - Flinders Medical Centre, Bedford Park
  - Royal Brisbane and Women's Hospital, Brisbane
  - Monash Medical Centre, Clayton
  - Concord Repatriation General Hospital, Concord
  - Fiona Stanley Hospital, Murdoch
- Canada (4):
  - University of Calgary Liver Unit, Calgary, Alberta
  - LMC Diabetes & Endocrinology Ltd, London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Nova Scotia Health Authority, Halifax
- France (6):
  - CHU Grenoble-Alpes - Hopital Michallon, La Tronche
  - Hôpital de la Croix Rousse - HCL, Lyon
  - CHU de Montpellier - Hopital Saint Eloi, Montpellier
  - AP-HP Hopital Saint Antoine, Paris
  - CHU Bordeaux - Hopital Haut-Leveque, Pessac
  - AP-HP Hopital Paul Brousse, Villejuif
- ID Clinic, Mysłowice, CET, Poland
- Fundacion de Investigacion (FDI), San Juan, Puerto Rico
- King's College Hospital, London, United Kingdom

REFERENCES:
- See also: EMMPACT Phase 2b Clinical Trial Homepage — https://www.emmpacttrial.com